CLINICAL TRIAL: NCT04609319
Title: ARIA: Real-world Utilization and Outcomes With Dacomitinib First-line Treatment for EGFR Mutation-positive Advanced Non-small Cell Lung Cancer Among Asian Patients - A Multi-center Chart Review
Brief Title: Real World Utilization and Outcomes With Dacomitinib First Line Treatment for EGFR Mutation-positive Advanced Non Small Cell Lung Cancer Among Asian Patients - A Multi Center Chart Review
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7471067
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — This is a non-interventional, real world study of Asian patients being treated with dacomitinib as first-line treatment for EGFR+ NSCLC

SUMMARY:
This is a longitudinal, consecutive case-series, multi-center study with mixed prospective and retrospective data collection. Data will be collected from eligible adults with EGFR mutation-positive advanced non-small cell lung cancer (NSCLC) treated with dacomitinib as first-line therapy from the date of advanced NSCLC diagnosis to the date of death, lost to follow-up, withdrawal of consent or end of study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥18 years) with histology-confirmed advanced NSCLC (TNM stage IIIB-IV);
* Presence of any EGFR-activating mutation (exon 19 deletion or exon 21 L858R substitution) or other uncommon EGFR mutations prior to anti-cancer treatment;
* Initiating dacomitinib as first-line treatment after confirmation of EGFR-mutation status (ie, no prior treatment with other EGFR TKI or systemic therapy);

Exclusion Criteria:

* Enrolled in any interventional clinical study or trial (however, patients enrolled in non-interventional, real world study may still be included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary cancer-treating hospitals in China, India and Malaysia are planned as participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - The First hospital of Jilin University, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Internal Medicine, Chinese Academy of Medical Sciences Cancer Hospital, Beijing
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning Province
- India (2):
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, DEL
  - Tata Memorial Center, Kolkata, Kolkata, West Bengal
- Malaysia (3):
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Beacon Hospital, Petaling Jaya

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wu L, Li J, Xu CR, Biswas B, Roy S, Tang KJ, Wang H, Liu Z, Batra U, Ho GF, Seng Hooi JL, Lu Y, Zhao M, Tho LM, Zhao J, He S, Huang J, Zhang H, Wong CH, Wu YL. Real-world use of and clinical outcomes with dacomitinib as first-line therapy in Asian patients with EGFR mutation-positive locally advanced or metastatic non-small cell lung cancer: Final analysis of the ARIA study. Lung Cancer. 2026 Jan;211:108856. doi: 10.1016/j.lungcan.2025.108856. Epub 2025 Nov 25. PMID 41365111
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants who were diagnosed with epidermal growth factor receptor (EGFR) mutation-positive advanced NSCLC and received first-line treatment with dacomitinib under routine clinical practice was included. Participants did not receive intervention as a part of this study. A total of 307 participants were enrolled. Of these, 8 participants were excluded from any analysis (7 participants failed to meet the eligibility criteria and 1 participant was a duplicate).
Pre-assignment Details: Data was collected retrospectively from medical records (1-Jan-2017 to 23-Nov-2021) or prospectively from prospective data collection (23-Nov-2021 to 28-May-2024) or mixed (retrospective and prospective, 1-Jan-2017 to 28-May-2024 [89 months]). Available data from eligible participants was evaluated in approximately 35.5 months (study start date: 11-June-2021 to study completion date: 28-May-2024) of this observational study as per its objectives.
Groups:
- Dacomitinib 30 mg: Participants who initiated treatment with dacomitinib as first line therapy at a dose of 30 milligrams (mg), once daily in a real world setting under routine clinical practice outside of clinical trials were included.
- Dacomitinib 45 mg: Participants who initiated treatment with dacomitinib as first line therapy at a dose of 45 mg, once daily in a real world setting under routine clinical practice outside of clinical trials were included.
- Dacomitinib Other Dose: Participants who initiated treatment with dacomitinib as first line therapy at a dose of 30 mg, twice daily or 15 mg, once daily in a real world setting under routine clinical practice outside of clinical trials were included.
Period: Overall Study
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Started (Eligible participants included in any analysis and this record.) | 159 | 138 | 2
Completed | 0 | 0 | 0
Not Completed | 159 | 138 | 2
Not completed — Death | 64 | 49 | 1
Not completed — Withdrawal of consent | 15 | 3 | 0
Not completed — Lost to Follow-up | 20 | 33 | 0
Not completed — Alive until end of follow-up | 60 | 53 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) included all eligible participants who fulfilled all inclusion and exclusion criteria and provided informed consent (or with institutional review board [IRB]/ independent ethics committee [IEC] waiver of informed consent).
Groups:
- Dacomitinib 30 mg: Participants who initiated treatment with dacomitinib as first line therapy at a dose of 30 mg, once daily in a real world setting under routine clinical practice outside of clinical trials were included.
- Total: Total of all reporting groups
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose | Total
Number analyzed (Participants) | 159 | 138 | 2 | 299
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (9.77) | 57.6 (9.29) | 70.5 (12.02) | 59.8 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 59 | 1 | 161
  Male | 58 | 79 | 1 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 145 | 125 | 2 | 272
  Malay | 1 | 0 | 0 | 1
  Indian | 12 | 13 | 0 | 25
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI): All Asian Participants
Description: BMI was derived from body weight and height, and it was calculated as weight divided by height^2.
Time Frame: Baseline (date of last non-missing measurement prior to dacomitinib initiation; from data collected for approx. [approximately] 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: FAS included all eligible participants who fulfilled all inclusion and exclusion criteria and provided informed consent (or with IRB/ IEC waiver of informed consent). Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilogram per square meter
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 96 | 114 | 1
Kilogram per square meter | 22.6 (3.57) | 23.1 (3.44) | 26.4

2. Primary Outcome: Number of Participants Classified According to Smoking Status: All Asian Participants
Description: Number of participants classified according to smoking status are presented in this outcome measure. Participants were classified into the following categories: current smoker, former smoker, never smoker and unknown.
Time Frame: Baseline (date of last non-missing measurement prior to dacomitinib initiation; from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: FAS included all eligible participants who fulfilled all inclusion and exclusion criteria and provided informed consent (or with IRB/ IEC waiver of informed consent).
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  Current smoker | 2 | 11 | 0
  Former smoker | 24 | 41 | 1
  Never smoker | 93 | 71 | 1
  Unknown | 40 | 15 | 0

3. Primary Outcome: Number of Participants Classified According to Comorbidities: All Asian Participants
Description: Number of participants classified According to comorbidities are presented in this outcome measure. Participants were classified into the following categories: any comorbidities, none and unknown.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  Any comorbidities | 44 | 22 | 1
  None | 97 | 109 | 1
  Unknown | 18 | 7 | 0

4. Primary Outcome: Number of Participants Classified According to NSCLC Staging: All Asian Participants
Description: The number of participants classified according to the disease stages as 3B, 3C, 4A and 4B were reported in this outcome measure. Cancer stages were classified based on tumor size (T), metastasis to regional lymph nodes (LN) [N] and distant metastasis (M). Stages were 3B, 3C, 4A and 4B. Stage 3B (T1N3M0, T2N3M0, T3N2M0, T4N2M0). Stage 3C (T3N3M0 and T4N3M0), Stage 4A (anyT, anyN and M1a/M1b), Stage 4B (anyT, anyN and M1c). where T1: <=3 cm; T2: >3 to <=5 cm; T3: >5 to <=7 cm; T4: >7cm. N0: not spread to regional LN; N1: spread to ipsilateral pulmonary or hilar nodes; N2: spread to ipsilateral mediastinal or subcarinal nodes; N3: spread to contralateral mediastinal, hilar, or supraclavicular nodes. M0: no distant metastasis; M1a: malignant pleural or pericardial effusion or pleural or pericardial nodules or separate tumor nodule(s) in a contralateral lobe; M1b: single extrathoracic metastasis; M1c= multiple extrathoracic metastases (1 or >1 organ).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  3B | 6 | 8 | 2
  3C | 0 | 4 | 0
  4A | 56 | 46 | 0
  4B | 97 | 80 | 0

5. Primary Outcome: Number of Participants Classified According to Eastern Cooperative Oncology Group (ECOG) Performance Status: All Asian Participants
Description: ECOG performance classified as: Grade 0: fully active, able to carry on all pre-disease performance without restriction; Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature; Grade 2: ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours; Grade 3: capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: completely disabled, cannot carry on selfcare and totally confined to bed or chair and Grade 5: dead. Higher score indicated worse health status.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  Grade 0 | 20 | 11 | 0
  Grade 1 | 59 | 80 | 0
  Grade 2 | 0 | 5 | 1
  Grade 3 | 2 | 1 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0
  Unknown | 73 | 40 | 1
  Missing | 5 | 1 | 0

6. Primary Outcome: Number of Participants Classified According to Type of EGFR Mutation: All Asian Participants
Description: Number of participants classified according to type of EGFR mutation were reported in this outcome measure. One participant may have more than one mutation. Participants were classified into the following rows: EGFR exon 19 deletion, EGFR exon 21 L858R substitution, EGFR T790M mutation and other.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  EGFR exon 19 deletion | 54 | 36 | 1
  EGFR exon 21 L858R substitution | 102 | 89 | 1
  EGFR T790M mutation | 0 | 2 | 0
  Other | 22 | 37 | 0

7. Primary Outcome: Number of Participants Classified According to Number of Oral Dose Modifications: All Asian Participants
Description: Number of participants with dacomitinib oral dose modification (any dose change) from initial dacomitinib therapy are presented in this outcome measure. Participants were classified into the following categories: no dose modification, one dose modification, two dose modifications and more than two dose modifications.
Time Frame: From start of dacomitinib treatment until discontinuation/end of treatment (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  No dose modification | 128 | 67 | 1
  One dose modification | 16 | 41 | 0
  Two dose modifications | 11 | 29 | 0
  More than two dose modifications | 4 | 1 | 1

8. Primary Outcome: Number of Participants Classified According to Number of Oral Dose Interruptions: All Asian Participants
Description: Number of participants with dacomitinib dose interruption (dacomitinib treatment being temporarily stopped) were reported in this outcome measure. Participants were classified into the following categories: no dose interruption, one dose interruption, two dose interruptions and more than two dose interruptions.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants
  No dose interruptions | 142 | 115 | 1
  One dose interruption | 10 | 20 | 0
  Two dose interruptions | 4 | 2 | 1
  More than two dose interruptions | 3 | 1 | 0

9. Primary Outcome: Number of Participants With Any Oral Dose Discontinuation: All Asian Participants
Description: Number of participants with dacomitinib dose discontinuation (dacomitinib treatment permanently stopped) were reported in this outcome measure.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants | 116 | 105 | 2

10. Primary Outcome: Duration of Dacomitinib Therapy: All Asian Participants
Description: Duration of dacomitinib therapy (dacomitinib last dose date - dacomitinib initiation date + 1 day) was reported in this outcome measure.
Time Frame: First dose of dacomitinib till discontinuation/ end of dacomitinib treatment (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Months | 17.4 [1.1 to 68.1] | 16.6 [0.7 to 48.9] | 14.9 [8.9 to 20.8]

11. Primary Outcome: Time To Treatment Failure (TTF): All Asian Participants
Description: TTF was defined as the time from date of dacomitinib initiation to date of dacomitinib permanent discontinuation (for any reason), first disease progression (PD), or death (from any cause), whichever came first. PD was defined as cancer worsening based on radiologist's interpretation of the imaging and/or clinician's assessment, and after initiation of first-line dacomitinib treatment. Participants who remained on dacomitinib without an event until end of follow-up were censored at the date of last known contact/visit date. Participants lost to follow-up were censored based on the last known contact/visit date. Kaplan-Meier method was used for analysis.
Time Frame: From dacomitinib treatment initiation to dacomitinib discontinuation, PD or death due to any cause, whichever came first or censoring date (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Months | 15.8 [13.40 to 19.88] | 17.7 [14.39 to 21.16] | 14.5 [8.34 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated due to insufficient number of participants with events.

12. Secondary Outcome: Progression-free Survival (PFS): All Asian Participants
Description: PFS was defined as date of dacomitinib initiation to date of first PD or death from any cause, whichever came first. PD was defined as cancer worsening based on radiologist's interpretation of the imaging and/or clinician's assessment, and after initiation of first-line dacomitinib treatment. Participants without PD and remained alive (i.e. no date of death) until end of follow-up were censored at the date of last known contact/visit date. Participants lost to follow-up were censored based on the last known contact/visit date. Kaplan-Meier method was used for analysis.
Time Frame: From dacomitinib treatment initiation to PD or death due to any cause, whichever came first or censoring date (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Months | 18.3 [15.47 to 26.51] | 21.0 [17.38 to 24.15] | 14.5 [8.34 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

13. Secondary Outcome: Number of Participants With Adverse Events (AEs): All Asian Participants
Description: AE was any untoward medical occurrence in a participant or clinical investigation participant administered sponsor's product and which did not necessarily have a causal relationship with the product.
Time Frame: From dacomitinib treatment initiation to death or end of study whichever occurred first (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 159 | 138 | 2
Participants | 79 | 82 | 1

14. Secondary Outcome: TTF: Chinese Participants With Common EGFR Mutation
Description: TTF was defined as the time from date of dacomitinib initiation to date of dacomitinib permanent discontinuation (for any reason), first PD, or death (from any cause), whichever came first. PD was defined as cancer worsening based on radiologist's interpretation of the imaging and/or clinician's assessment, and after initiation of first-line dacomitinib treatment. Participants who remained on dacomitinib without an event until end of follow-up were censored at the date of last known contact/visit date. Participants lost to follow-up were censored based on the last known contact/visit date. Kaplan-Meier method was used for analysis.
Time Frame: as for outcome 11
Population: FAS included all eligible participants who fulfilled all inclusion and exclusion criteria and provided informed consent (or with IRB/ IEC waiver of informed consent). Here, "Overall Number of Participants Analyzed" signifies Chinese participants with common EGFR mutation evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 133 | 113 | 1
Months | 17.3 [14.46 to 20.60] | 18.9 [14.52 to 22.51] | NA [NA to NA] — There was only 1 participant evaluable with TTF of 8.3 months.

15. Secondary Outcome: PFS: Chinese Participants With Common EGFR Mutation
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 133 | 113 | 1
Months | 20.3 [16.99 to 30.29] | 21.2 [18.40 to 25.33] | NA [NA to NA] — There was only 1 participant evaluable with PFS of 8.3 months.

16. Secondary Outcome: Number of Participants With AEs: Chinese Participants With Common EGFR Mutation
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 133 | 113 | 1
Participants | 60 | 67 | 0

17. Secondary Outcome: Number of Participants Classified According to Starting Dose of Dacomitinib as First-line Therapy: Chinese Participants With Common EGFR Mutation
Description: Number of participants classified according to starting dose of dacomitinib (30 mg, 45 mg or other dose) as first-line in Chinese participants with common EGFR mutations are presented in this outcome measure.
Time Frame: as for outcome 7
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 133 | 113 | 1
Participants
  30 mg once daily | 133 | 0 | 0
  45 mg once daily | 0 | 113 | 0
  Other dose | 0 | 0 | 1

18. Secondary Outcome: Number of Participants Without Oral Dose Modifications: Chinese Participants With Common EGFR Mutation
Description: Number of participants without any dacomitinib dose modification (any dose change) from initial dacomitinib therapy in Chinese participants with common EGFR mutations are presented in this outcome measure.
Time Frame: as for outcome 7
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
Number analyzed (Participants) | 133 | 113 | 1
Participants | 111 | 55 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality: From dacomitinib treatment initiation to death or end of study whichever occurred first (from data collected for approx. 89 months); data was evaluated in this observational study for approx. 35.5 months; for adverse events it was not applicable due to non-interventional nature of the study adverse events were not planned to be assessed/monitored
Description: Due to non-interventional nature of the study, adverse events and their seriousness were not monitored/assessed which explains at risk as zero.
Arm/Group | Dacomitinib 30 mg | Dacomitinib 45 mg | Dacomitinib Other Dose
All-Cause Mortality (participants affected / at risk) | 64/159 | 49/138 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to non-interventional nature of the study, adverse events and their seriousness were not monitored/assessed; only summarized data is reported per objectives of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT04609319/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04609319/SAP_001.pdf